CLINICAL TRIAL: NCT03692390
Title: A Pragmatic Randomized Controlled Trial of Virtual Reality vs. Standard-of-Care for Comfort Before and After Sedation in the Emergency Department
Brief Title: Virtual Reality vs. Standard-of-Care for Comfort Before and After Sedation in the Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ran Goldman, Professor and Co-head of the Division of Clinical Pharmacology, Division of Emergency Medicine, Department of Pediatrics; Investigator, BC Children's Hospital, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H18-01949
Record Dates: First submitted 2018-09-20; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Procedural Sedation
Keywords: Virtual Reality; Heart Rate; Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Participants are distracted by wearing the virtual reality headset and watching a roller coaster app while undergoing procedural sedation
  Interventions: Device: Virtual Reality
- Standard-of-Care (No Intervention): Participants are distracted with Standard-of-Care by doctors, nurses, nurse practitioners, child life specialists and/or parents.

INTERVENTIONS:
Device: Virtual Reality — Participants wear a Virtual Reality headset that consists of a ASUS phone and a VOX+ Z3 3D Virtual Reality Headset. The phone runs the VR Roller Coaster app to produce the virtual environment.
  Arms: Virtual Reality

SUMMARY:
Children often need procedural sedation in the emergency department during painful procedures (such as reducing fractures).

Virtual Reality (VR) is an immersive experience using sight, sound, and position sense. Using VR may enhance distraction during the painful procedure and may reduce attention to pain. VR may also reduce anxiety during sedation induction by reducing providing an alternative stimulus.

This study will randomize children (6 - 16 years old) to receive Virtual Reality or standard of care while undergoing procedural sedation. Investigators will measure heart rate, blood pressure, satisfaction (child, parent, provider), amount of sedatives used and compare between the two groups.

ELIGIBILITY:
INCLUSION CRITERIA

1. Children age 6 to 16 years
2. The managing physician determines need for procedural sedation
3. Parents will sign a consent form and children will sign an assent form

EXCLUSION CRITERIA

1. Children with conditions that may prohibit participation or evaluation of the procedure (such as developmental delay, autism, inability to communicate)
2. Triage category 1 (resuscitation)
3. Facial features or injury prohibiting wearing the VR goggles

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-09-21 (Estimated); Study Completion 2019-09-21 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate as measured by heart rate monitor | During the procedure at 1 minute intervals
  The heart rate monitor will consistently display participant heart rate. Heart rate will be recorded at 1 minute intervals. The difference in heart rate from recommended mean heart rate based on age will be calculated and compared between groups.
Change in Blood Pressure as measured by blood pressure monitor | During the procedure at 1 minute intervals
  The blood pressure monitor will display participant blood pressure. Blood pressure will be recorded at 1 minute intervals. The difference in blood pressure from recommended mean blood pressure (systolic and diastolic) based on age will be calculated and compared between groups.

SECONDARY OUTCOMES:
Emergence Phenomenon as measured by yes/no questions regarding participant experience. | Immediately after the procedure and by phone the next day
  Patients will be asked whether they experienced nightmares, day-dreaming, or feeling unwell. Number of patients who experienced these negative emergence phenomenon will be tabulated and compared across groups.
Satisfaction among Children by global rating scale | Immediately after the procedure
  Children will be asked "On a scale of 0-10, how did the procedure go?" A score of 0 represents not very well and a score of 10 represents very well.
Satisfaction among Guardians by global rating scale | Immediately after the procedure
  Guardians will be asked "On a scale of 0-10, how did the procedure go?" A score of 0 represents not very well and a score of 10 represents very well.
Satisfaction among Emergency Staff by global rating scale | Immediately after the procedure
  Emergency Staff will be asked "How satisfied are you with how the procedure went?" A score of 0 represents not very well and a score of 10 represents very well.
Type and dose of medication | Intraoperative
  Amount of medication and what medications were used will be gathered from the nursing notes.
Time difference of the procedure | Intraoperative
  Time the procedure takes to complete with or without VR will be recorded to determine if there is any difference.
Length of stay in the Emergency Department | Intraoperative
  Length of stay in the Emergency Department will also be recorded. This will be determined by the intake time noted by triage and the discharge time as witnessed by research assistant or, if unseen, by the time noted on the discharge paperwork.

CONTACTS AND LOCATIONS:
Overall Officials: Ran Goldman, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada